CLINICAL TRIAL: NCT04782583
Title: Shifting of Intrauterine Device and Use of the Menstrual Cup: Case-control Study
Acronym: CUP-DIU
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: HPD_2019_18
Record Dates: First submitted 2021-01-13; First posted 2021-03-04 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Menstrual Cup; Intrauterine Device Migration
MeSH Terms: conditions — Intrauterine Device Migration | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CAS
  Interventions: Other: Questionnaire
- TEMOIN
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — questionnaire for the patients and the volontaire

SUMMARY:
In France, 26% of women of childbearing age use an intrauterine device (IUD) containing copper or levonorgestrel as a method of contraception. Failures of IUD contraception are mainly due to shifting or expulsion of the IUD. The risk factors for expulsion of IUDs most often found in the literature are young age (<25 years), the existence of menorrhagia, dysmenorrhea, being a carrier of a copper IUD rather than a levonorgestrel IUD , a history of IUD expulsion, nulliparity, and an anomaly of the uterine cavity unrecognized (fibroma, adenomyosis).

More and more women are turning to menstrual cups (MCs) as a means of periodic protection. But the use of MC has also been mentioned as a risk factor for IUD expulsion (via a suction effect). In May 2013, reports of displacement, rupture, or even expulsion of copper IUDs in CM users were reported to ANSM.

However, few studies have examined the risks associated with the concomitant use of an MC and an IUD. The data are contradictory and insufficient to provide a clear answer to women. Hence the interest in carrying out a larger prospective study to explore the relationship between IUD expulsion and the use of MC.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over
* Consultant for one of the following reasons:

  * IUD control
  * IUD expulsion
  * Pregnancy on IUD
  * Other reason that required an ultrasound for the IUD
* Consent to participate in the study

Exclusion Criteria:

* Patient benefiting from a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an intrauterine device for contraception.
Sampling Method: Non-Probability Sample
Enrollment: 740 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Evaluating the risk of IUD displacement in patients using menstrual cup | 1 DAY
  Transvaginal ultrasounds will be used to monitor the position of the intrauterine device in patients using a menstrual cup.

CONTACTS AND LOCATIONS:
Locations (1):
- cabinet IPSO, Paris, France

REFERENCES:
- [Derived] Claire J, Mir S, Dumortier I, Liard R, Yavchitz A, Le Cossec C, Picard H. The use of a menstrual cup as a risk factor for displacement of intrauterine devices: a case-control study. Contracept Reprod Med. 2025 May 6;10(1):33. doi: 10.1186/s40834-025-00366-3. PMID 40329407